CLINICAL TRIAL: NCT00099853
Title: Efficacy and Safety of Vildagliptin in Combination With Pioglitazone in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A2304
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Vildagliptin 50 mg qd + pioglitazone 45 mg qd (Experimental): Vildagliptin 50 mg qd + pioglitazone 45 mg qd for 24 weeks
  Interventions: Drug: Vildagliptin; Drug: pioglitazone
- Vildagliptin 50 mg bid + pioglitazone 45 mg qd (Experimental): Vildagliptin 50 mg bid + pioglitazone 45 mg qd for 24 weeks
  Interventions: Drug: Vildagliptin; Drug: pioglitazone
- Vildagliptin placebo + pioglitazone 45 mg qd (Placebo Comparator): Vildagliptin placebo + pioglitazone 45 mg qd for 24 weeks
  Interventions: Drug: pioglitazone; Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin 50 mg tablets
  Other Names: LAF237; Galvus
  Arms: Vildagliptin 50 mg bid + pioglitazone 45 mg qd; Vildagliptin 50 mg qd + pioglitazone 45 mg qd
Drug: pioglitazone — pioglitazone 45 mg qd
Drug: Placebo — Vildagliptin matching placebo
  Arms: Vildagliptin placebo + pioglitazone 45 mg qd

SUMMARY:
Many people with type 2 diabetes cannot maintain target blood glucose levels when taking a single oral drug. The purpose of this study is to assess the safety and effectiveness of vildagliptin, an unapproved drug, in lowering overall blood glucose levels when added to pioglitazone in people with type 2 diabetes not at target blood glucose levels on either pioglitazone or rosiglitazone alone.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose criteria must be met
* Previously responded, as defined by the protocol, to treatment with pioglitazone or rosiglitazone
* Body mass index (BMI) in the range 22-45

Exclusion Criteria:

* Type 1 diabetes
* Pregnancy or lactation
* Evidence of serious cardiovascular complications
* Evidence of serious diabetic complications
* Laboratory value abnormalities as defined by the protocol
* Known sensitivity to pioglitazone
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2004-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c after 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose at 24 weeks
Patients with endpoint HbA1c <7% after 24 weeks
Patients with reduction in HbA1c >/= to 0.7% after 24 weeks
Adverse event profile after 24 weeks of treatment
Change from baseline in HbA1c at 24 weeks for patients with high baseline HbA1c vs low baseline HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Garber AJ, Schweizer A, Baron MA, Rochotte E, Dejager S. Vildagliptin in combination with pioglitazone improves glycaemic control in patients with type 2 diabetes failing thiazolidinedione monotherapy: a randomized, placebo-controlled study. Diabetes Obes Metab. 2007 Mar;9(2):166-74. doi: 10.1111/j.1463-1326.2006.00684.x. PMID 17300592
- See also: Results for CLAF237A2304 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2286